CLINICAL TRIAL: NCT05214573
Title: Second-line Therapies for Patients With Type 2 Diabetes and Moderate Cardiovascular Disease Risk
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Rozalina G. McCoy, Principal Investigator, Mayo Clinic
Other Study IDs: 21-007688
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Cardiac Disease
Keywords: Diabetes; Type 2 diabetes; Cardiovascular disease; Comparative effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases; Diabetes Mellitus; Cardiovascular Diseases | interventions — Sodium-Glucose Transporter 2 Inhibitors; Dipeptidyl-Peptidase IV Inhibitors; Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aims 1, 2B, and 3 Groups: De-identified administrative claims with linked laboratory results, electronic health record (EHR), and mortality data from the OptumLabs Data Warehouse (OLDW) and Medicare fee-for-service data (Medicare parts A, B, D) will be utilized to identify adults (≥21 years) with T2D (established using validated Healthcare Effectiveness Data and Information Set criteria) who first filled any study drug GLP-1RA, SGLT2i, DPP-4i, or SU between 1/1/2014-12/31/2021. This arm was exempt from Mayo Clinic Institutional Review Board review and informed consent requirements were not applicable as this arm used deidentified administrative claims data.
  Interventions: Drug: Glucagon like peptide 1 receptor agonist; Drug: Sodium-glucose cotransporter 2 inhibitor; Drug: Dipeptidyl Peptidase 4 Inhibitor; Drug: Sulfonylurea
- Aim 2A Group: Adults with Type 2 diabetes treated with one or more of the study medications (GLP-1RA, SGLT2i, DPP-4i, or SU) and not treated with insulin who receive medical care at Mayo Clinic Rochester or Mayo Clinic Health System in Minnesota or Wisconsin. This arm was not exempt from Mayo Clinic Institutional Review Board review and informed consent requirements were applicable as this arm collected prospective data.

INTERVENTIONS:
Drug: Glucagon like peptide 1 receptor agonist — Patients in the data who filled a glucagon-like peptide-1 receptor agonist medication
  Groups: Aims 1, 2B, and 3 Groups
Drug: Sodium-glucose cotransporter 2 inhibitor — Patients in the data who filled a sodium-glucose cotransporter 2 inhibitor
  Groups: Aims 1, 2B, and 3 Groups
Drug: Dipeptidyl Peptidase 4 Inhibitor — Patients in the data who filled a dipeptidyl peptidase-4 inhibitor
  Groups: Aims 1, 2B, and 3 Groups
Drug: Sulfonylurea — Patients in the data who filled a sulfonylurea
  Groups: Aims 1, 2B, and 3 Groups

SUMMARY:
We will use the target trial framework for causal inference to conduct this observational retrospective cohort study that uses claims data of adults with type 2 diabetes (T2D) included in the de-identified datasets of OptumLabs Data Warehouse (OLDW) and Medicare fee-for-service.

In Aim 1, we will emulate a target trial comparing the effectiveness of glucagon-like peptide-1 receptor agonists (GLP-1RA), sodium-glucose cotransporter 2 inhibitors (SGLT2i), dipeptidyl peptidase-4 inhibitors (DPP-4i), and sulfonylureas (SU) in adults with T2D at moderate risk of cardiovascular disease (CVD) with regard to major adverse cardiovascular events (MACE), expanded MACE, microvascular complications, severe hypoglycemia, and other adverse events.

In Aim 2, we will compare these four drug classes in the same population of adults with T2D included in OLDW and Medicare fee-for-service data with respect to a set of composite outcomes identified by a group of patients with T2D as being most important to them. Specifically, in Aim 2A, we will prospectively elicit patient preferences toward various treatment outcomes (e.g., hospitalization, kidney disease) using a participatory ranking exercise, then use these rankings to generate individually weighted composite outcomes. Then, in Aim 2B, we will estimate patient-centered treatment effects of four different second-line T2D medications that reflect the patient's value for each outcome.

In Aim 3, we will compare different medications within each of the four therapeutic classes with respect to MACE.

DETAILED DESCRIPTION:
Study Design: We will use the target trial framework for causal inference to conduct this observational cohort study.

Comparators: Aims 1-2 compare the GLP-1RA, SGLT2i, DPP-4i, and SU classes, while Aim 3 compares the individual drugs within each therapeutic class.

Population: Using data from OptumLabs Data Warehouse linked to 100% Medicare FFS claims, we will identify adults (≥21 years) with T2D at moderate risk for CVD who started a GLP-1RA, SGLT2i, DPP-4i, or SU

Outcomes: In AIMs 1 and 3, the primary outcome will be time to MACE (non-fatal MI, non-fatal stroke, all-cause mortality). Secondary outcomes will include times to expanded MACE (MACE, HF hospitalizations, revascularization procedures) and its components, lower extremity complications, severe hypoglycemia, microvascular complications, and other significant adverse events. In AIM 2A, we will elicit patient preferences toward various treatment outcomes using a participatory ranking exercise, use these rankings to generate individually weighted composite outcomes, and then estimate patient-centered treatment effects of GLP-1RA, SGLT2i, DPP4i, and SU reflecting the patient values for each of the outcomes.

Timeframe: January 1, 2014 to December 31, 2021.

Methods: Inverse probability weighting will be used to emulate baseline randomization for pairwise comparisons between the drug classes (AIMs 1-2) and individual drugs within each class (AIM 3). Causal cumulative incidence rates will be estimated in the weighted sample using the targeted maximum likelihood estimator adjusting for time-dependent confounding and loss-to-follow-up.

ELIGIBILITY:
Inclusion Criteria for all Aims

* ≥ 21 years old.
* Diagnosis of Type 2 diabetes.
* Use of ≥ 1 study drug (GLP-1RA, SGLT2i, DPP-4i, SU).

Exclusion Criteria for Aims 1, 2B, 3

* Fill for any study drug during the baseline period or simultaneous (within 30 days) start of ≥2 study drugs
* Insulin use
* Type 1 diabetes
* High risk of CVD
* Pregnancy
* Metastatic cancer

Exclusion Criteria for Aim 2A

* Insulin use.
* Cognitive impairment.
* Terminal or advanced illness.
* Non-English speaking.
* Residency in a long-term care setting.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aims 1, 2B, 3: De-identified data sets using laboratory results, electronic health record and mortality data from the OptumLabs Data Warehouse (OLDW) and Medicare fee-for-service data.
  Aim 2A: Adults with Type 2 diabetes receiving care from primary care and endocrinology practices in Mayo Clinic Rochester, MN or Mayo Clinic Health System in Minnesota and Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 386301 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozalina McCoy, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Neumiller JJ, Herrin J, Swarna KS, Polley EC, Galindo RJ, Umpierrez GE, Deng Y, Ross JS, Mickelson MM, McCoy RG. Kidney Outcomes with Glucagon-Like Peptide-1 Receptor Agonists, Sodium-Glucose Cotransporter 2 Inhibitors, Dipeptidyl Peptidase-4 Inhibitors, and Sulfonylureas in Type 2 Diabetes and Moderate Cardiovascular Risk. Clin J Am Soc Nephrol. 2024 Oct 8;20(2):206-17. doi: 10.2215/CJN.0000000587. Online ahead of print. PMID 39729347
- [Derived] McCoy RG, Herrin J, Swarna KS, Deng Y, Kent DM, Ross JS, Umpierrez GE, Galindo RJ, Crown WH, Borah BJ, Montori VM, Brito JP, Neumiller JJ, Mickelson MM, Polley EC. Effectiveness of glucose-lowering medications on cardiovascular outcomes in patients with type 2 diabetes at moderate cardiovascular risk. Nat Cardiovasc Res. 2024 Apr;3(4):431-440. doi: 10.1038/s44161-024-00453-9. Epub 2024 Apr 3. PMID 38846711
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in the arm "Aims 1, 2B, and 3 groups", were considered enrolled in the trial even though this arm was exempt from Mayo Clinic Institutional Review Board review and informed consent requirements were not applicable as this arm used deidentified administrative claims data.
Groups:
- Aims 1, 2B, and 3 Groups: De-identified administrative claims with linked laboratory results, electronic health record (EHR), and mortality data from the OptumLabs Data Warehouse (OLDW) and Medicare fee-for-service data (Medicare parts A, B, D) were utilized to identify adults (≥21 years) with T2D (established using validated Healthcare Effectiveness Data and Information Set criteria) who first filled any study drug GLP-1RA, SGLT2i, DPP-4i, or SU between 1/1/2014-12/31/2021. The arm was exempt from Mayo Clinic Institutional Review Board review and informed consent requirements were not applicable as this arm used deidentified administrative claims data.
  Glucagon like peptide 1 receptor agonist: Patients in the data who filled a glucagon-like peptide-1 receptor agonist medication
  Sodium-glucose cotransporter 2 inhibitor: Patients in the data who filled a sodium-glucose cotransporter 2 inhibitor
  Dipeptidyl Peptidase 4 Inhibitor: Patients in the data who filled a dipeptidyl peptidase-4 inhibitor
  Sulfonylurea: Patients in the data who filled a sulfonylurea
- Aim 2A Group: Adults with Type 2 diabetes treated with one or more of the study medications (GLP-1RA, SGLT2i, DPP-4i, or SU) and not treated with insulin who received medical care at Mayo Clinic Rochester or Mayo Clinic Health System in Minnesota or Wisconsin. This arm was not exempt from Mayo Clinic Institutional Review Board review and informed consent requirements were applicable as this arm collected prospective data.
Period: Overall Study
Arm/Group | Aims 1, 2B, and 3 Groups | Aim 2A Group
Started | 386276 | 25
Completed | 380352 | 25
Not Completed | 5924 | 0
Not completed — Physician Decision | 5924 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aims 1, 2B, and 3 Groups | Aim 2A Group | Total
Number analyzed (Participants) | 386276 | 25 | 386301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 131786 | 19 | 131805
  >=65 years | 254490 | 6 | 254496
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190394 | 13 | 190407
  Male | 195882 | 12 | 195894
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33165 | 5 | 33170
  Not Hispanic or Latino | 341028 | 19 | 341047
  Unknown or Not Reported | 12083 | 1 | 12084
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10982 | 0 | 10982
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39454 | 1 | 39455
  White | 285574 | 20 | 285594
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 50266 | 4 | 50270
Region of Enrollment [Number; unit: participants]
  United States | 386276 | 25 | 386301

OUTCOME MEASURES:

1. Primary Outcome: 3-point Major Adverse Cardiovascular Event (MACE)
Description: The probability of 3-point MACEs experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylureas (SU) defined as non-fatal myocardial infarction (MI), non-fatal stroke, and mortality. The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: 380352 total participants were analyzed. Those 380352 participants were further broken down into the following categories DPP4i (82438), GLP-1RA (44255), SGLT2i (46473), Sulfonylureas (SU) (207186), respectively.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 380352
Hazard Ratio
  GLP-1RA versus DPP4i: number analyzed (Participants) | 126693
  GLP-1RA versus DPP4i | 0.87 [0.82 to 0.93]
  SGLT2i versus DPP4i: number analyzed (Participants) | 128911
  SGLT2i versus DPP4i | 0.85 [0.81 to 0.90]
  SU versus DPP4i: number analyzed (Participants) | 289624
  SU versus DPP4i | 1.19 [1.16 to 1.22]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 90728
  SGLT2i versus GLP-1RA | 0.97 [0.90 to 1.05]
  SU versus GLP-1RA: number analyzed (Participants) | 251441
  SU versus GLP-1RA | 1.36 [1.28 to 1.46]
  SU versus SGLT2i: number analyzed (Participants) | 253659
  SU versus SGLT2i | 1.40 [1.33 to 1.47]

2. Primary Outcome: Expanded Major Adverse Cardiovascular Events (MACE) and Its Components
Description: The probability of 3-point MACEs (non-fatal MI, non-fatal stroke, mortality) plus heart failure hospitalization and revascularization procedure events experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylureas (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 380352
Hazard Ratio
  GLP-1RA versus DPP4i: number analyzed (Participants) | 126693
  GLP-1RA versus DPP4i | 0.95 [0.91 to 1.00]
  SGLT2i versus DPP4i: number analyzed (Participants) | 128911
  SGLT2i versus DPP4i | 0.93 [0.89 to 0.96]
  SU versus DPP4i: number analyzed (Participants) | 289624
  SU versus DPP4i | 1.14 [1.12 to 1.17]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 90728
  SGLT2i versus GLP-1RA | 0.97 [0.92 to 1.02]
  SU versus GLP-1RA: number analyzed (Participants) | 251441
  SU versus GLP-1RA | 1.20 [1.15 to 1.26]
  SU versus SGLT2i: number analyzed (Participants) | 253659
  SU versus SGLT2i | 1.24 [1.20 to 1.28]

3. Primary Outcome: Patient Preferences for Second-line Type 2 Diabetes Medication Treatment Outcomes
Description: Patients ranked treatment outcomes using a participatory ranking questionnaire. The questionnaire included a list of 16 health outcomes and eight medication attributes, with opportunities for participants to add outcomes and attributes into the ranking lists. During the exercise, participants were asked to assign each outcome and attribute to one of three mutually exclusive categories: "very important," "somewhat important," or "not very important," based on the degree to which each outcome or attribute would influence their choice of medication. Results shown below reflect the health outcomes/medication attributes that were ranked "very important" by patients.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 2A Group
Number analyzed (Participants) | 25
Participants
  Serious Infection | 2
  Being admitted | 2
  Pancreatitis | 3
  Issues with your feet | 4
  Eye Issues | 4
  Worsening Kidney Function | 4
  Very low blood sugar | 4
  Cancer | 7
  Vessel Blockages | 7
  Stroke | 7
  Amputation | 10
  Heart Attack | 10
  End Stage Kidney Disease (ESKD) | 11
  Death | 12
  Heart Failure | 13
  Blindness | 16

4. Secondary Outcome: Non-fatal Myocardial Infarction (MI)
Description: The probability of a non-fatal MI experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylureas (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 380352
Hazard Ratio
  GLP-1RA versus DPP4i: number analyzed (Participants) | 126693
  GLP-1RA versus DPP4i | 0.89 [0.78 to 1.01]
  SGLT2i versus DPP4i: number analyzed (Participants) | 128911
  SGLT2i versus DPP4i | 0.93 [0.85 to 1.02]
  SU versus DPP4i: number analyzed (Participants) | 289624
  SU versus DPP4i | 1.21 [1.15 to 1.26]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 90728
  SGLT2i versus GLP-1RA | 1.05 [0.91 to 1.21]
  SU versus GLP-1RA: number analyzed (Participants) | 251441
  SU versus GLP-1RA | 1.35 [1.20 to 1.53]
  SU versus SGLT2i: number analyzed (Participants) | 253659
  SU versus SGLT2i | 1.30 [1.19 to 1.41]

5. Secondary Outcome: Non-fatal Stroke Events
Description: The probability of non-fatal stroke events experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylureas (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 380352
Hazard Ratio
  GLP-1RA versus DPP4i: number analyzed (Participants) | 126693
  GLP-1RA versus DPP4i | 0.89 [0.78 to 1.02]
  SGLT2i versus DPP4i: number analyzed (Participants) | 128911
  SGLT2i versus DPP4i | 0.89 [0.81 to 0.98]
  SU versus DPP4i: number analyzed (Participants) | 289624
  SU versus DPP4i | 1.18 [1.13 to 1.24]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 90728
  SGLT2i versus GLP-1RA | 1.00 [0.86 to 1.16]
  SU versus GLP-1RA: number analyzed (Participants) | 251441
  SU versus GLP-1RA | 1.33 [1.17 to 1.50]
  SU versus SGLT2i: number analyzed (Participants) | 253659
  SU versus SGLT2i | 1.33 [1.22 to 1.45]

6. Secondary Outcome: All-cause Mortality
Description: The probability of all-cause mortality events experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, Sulfonylureas (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 380352
Hazard Ratio
  GLP-1RA versus DPP4i: number analyzed (Participants) | 126693
  GLP-1RA versus DPP4i | 0.86 [0.78 to 0.94]
  SGLT2i versus DPP4i: number analyzed (Participants) | 128911
  SGLT2i versus DPP4i | 0.79 [0.73 to 0.85]
  SU versus DPP4i: number analyzed (Participants) | 289624
  SU versus DPP4i | 1.22 [1.18 to 1.26]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 90728
  SGLT2i versus GLP-1RA | 0.92 [0.82 to 1.03]
  SU versus GLP-1RA: number analyzed (Participants) | 251441
  SU versus GLP-1RA | 1.42 [1.30 to 1.56]
  SU versus SGLT2i: number analyzed (Participants) | 253659
  SU versus SGLT2i | 1.55 [1.44 to 1.66]

7. Secondary Outcome: Severe Hypoglycemia
Description: The probability of emergency department visits or hospitalization for hypoglycemia experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylurea (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 380352
Hazard Ratio
  GLP-1RA versus DPP4i: number analyzed (Participants) | 126693
  GLP-1RA versus DPP4i | 0.63 [0.51 to 0.76]
  SGLT2i versus DPP4i: number analyzed (Participants) | 128911
  SGLT2i versus DPP4i | 0.56 [0.46 to 0.68]
  SU versus DPP4i: number analyzed (Participants) | 289624
  SU versus DPP4i | 2.51 [2.29 to 2.75]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 90728
  SGLT2i versus GLP-1RA | 0.90 [0.70 to 1.16]
  SU versus GLP-1RA: number analyzed (Participants) | 251441
  SU versus GLP-1RA | 4.00 [3.32 to 4.85]
  SU versus SGLT2i: number analyzed (Participants) | 253659
  SU versus SGLT2i | 4.46 [3.73 to 5.32]

8. Secondary Outcome: Incident End-stage Kidney Disease
Description: The probability of a new diagnosis of stage 5 or end-stage kidney disease experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylurea (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: 367452 total participants were analyzed. Those 367452 participants were further broken down into the following categories DPP4i (77042), GLP-1RA (42009), SGLT2i (53435), Sulfonylureas (SU) (194966), respectively.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 367452
Hazard Ratio
  SGLT2i versus DPP4i: number analyzed (Participants) | 130477
  SGLT2i versus DPP4i | 0.65 [0.56 to 0.76]
  GLP-1RA versus DPP4i: number analyzed (Participants) | 119051
  GLP-1RA versus DPP4i | 0.81 [0.66 to 0.99]
  SU versus DPP4i: number analyzed (Participants) | 272008
  SU versus DPP4i | 1.01 [0.93 to 1.08]
  SGLT2i versus SU: number analyzed (Participants) | 248401
  SGLT2i versus SU | 0.65 [0.56 to 0.75]
  GLP-1RA versus SU: number analyzed (Participants) | 236975
  GLP-1RA versus SU | 0.80 [0.66 to 0.97]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 95444
  SGLT2i versus GLP-1RA | 0.81 [0.64 to 1.02]

9. Secondary Outcome: Treatment for Diabetic Retinopathy or Macular Edema
Description: The probability of treatment for diabetic retinopathy and/or macular edema experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylurea (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: 371698 total participants were analyzed. Those 371698 participants were further broken down into the following categories DPP4i (78444), GLP-1RA (42265), SGLT2i (53476), Sulfonylureas (SU) (197513), respectively.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 371698
Hazard Ratio
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 95741
  SGLT2i versus GLP-1RA | 0.73 [0.55 to 0.97]
  SGLT2i versus DPP4i: number analyzed (Participants) | 131920
  SGLT2i versus DPP4i | 0.79 [0.64 to 0.97]
  SGLT2i versus SU: number analyzed (Participants) | 250989
  SGLT2i versus SU | 0.61 [0.50 to 0.74]
  GLP-1RA versus DPP4i: number analyzed (Participants) | 120709
  GLP-1RA versus DPP4i | 1.07 [0.85 to 1.35]
  GLP-1RA versus SU: number analyzed (Participants) | 239778
  GLP-1RA versus SU | 0.83 [0.67 to 1.03]
  SU versus DPP4i: number analyzed (Participants) | 275957
  SU versus DPP4i | 1.29 [1.17 to 1.42]

10. Secondary Outcome: Lower Extremity Complications
Description: The probability of foot and/or leg amputation, osteomyelitis, ulcer, abscess or Charcot arthropathy experienced by subjects treated with DPP4i, GLP-1RA, SGLT2i, or Sulfonylurea (SU). The probability was calculated and reported as the hazard ratio.
Time Frame: Retrospective Data between 1/1/2014 - 12/31/2022, up to 8 years, collected over a 2-year period
Population: 384451 total participants were analyzed. Those 384451 participants were further broken down into the following categories DPP4i (83937), GLP-1RA (43947), SGLT2i (46926), Sulfonylureas (SU) (209641), respectively.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Aims 1, 2B, and 3 Groups
Number analyzed (Participants) | 384451
Hazard Ratio
  SU versus DPP4i: number analyzed (Participants) | 293578
  SU versus DPP4i | 1.15 [1.11 to 1.19]
  SU versus GLP-1RA: number analyzed (Participants) | 253588
  SU versus GLP-1RA | 1.20 [1.13 to 1.28]
  SU versus SGLT2i: number analyzed (Participants) | 256567
  SU versus SGLT2i | 1.08 [1.02 to 1.14]
  SGLT2i versus GLP-1RA: number analyzed (Participants) | 90873
  SGLT2i versus GLP-1RA | 1.11 [1.03 to 1.21]
  GLP-1RA versus DPP4i: number analyzed (Participants) | 127884
  GLP-1RA versus DPP4i | 0.96 [0.89 to 1.02]
  SGLT2i versus DPP4i: number analyzed (Participants) | 130863
  SGLT2i versus DPP4i | 1.07 [1.00 to 1.13]

ADVERSE EVENTS:
Time Frame: Aims 1, 2B, and 3 Groups: Adverse events were collected from the time of first observed use of one of the four study medications (DPP4i, GLP-1RA, SGLT2i, Sulfonylurea) during the study period until either the end of the study, disenrollment from insurance plans in our database, or death (approximately 8 years), retrospective data collected over a 2-year period. Aim 2A Group: Adverse events were collected from the time of informed consent through study completion, approximately 1 hour.
Description: Aims 1, 2B, and 3 Groups: Adverse events were collected through de-identified administrative claims with linked laboratory results, electronic health record (EHR), and mortality data from the OptumLabs Data Warehouse (OLDW) and Medicare fee-for-service data (Medicare parts A, B, D). Aims 2A Group: Adverse events were collected through patient interviews.
Arm/Group | Aims 1, 2B, and 3 Groups | Aim 2A Group
All-Cause Mortality (participants affected / at risk) | 22208/386276 | 0/25
Serious Adverse Events (participants affected / at risk) | 40642/386276 | 0/25
Other Adverse Events (participants affected / at risk) | 62982/386276 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aims 1, 2B, and 3 Groups (N=386276) | Aim 2A Group (N=25)
Acute MI (Cardiac disorders) | 11372 | 0
Acute Stroke (Nervous system disorders) | 10647 | 0
Heart Failure Hospitalization (Cardiac disorders) | 10455 | 0
Chronic Kidney Disease Stage 5 or ESKD (Renal and urinary disorders) | 9216 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 4282 | NA
Amputation (Injury, poisoning and procedural complications) | 4661 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aims 1, 2B, and 3 Groups (N=386276) | Aim 2A Group (N=25)
Revascularization Procedure (Cardiac disorders) | 42514 | 0
Lower Extremity Complication (Injury, poisoning and procedural complications) | 21466 | 0
Treatment for Retinopathy (Eye disorders) | 4934 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT05214573/Prot_SAP_000.pdf